CLINICAL TRIAL: NCT03324204
Title: Shock Wave Therapy Versus Neuromuscular Training in Women With Patellofemoral Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Piotr Michalik, Principal Investigator, Medical University of Silesia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: kolanostudentki
Record Dates: First submitted 2017-07-18; First posted 2017-10-27 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Patellofemoral Pain Syndrome; Knee Pain Chronic
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular Training (Experimental): Each session lasted 30 minutes and consisted of three sets of exercises with 20-30 repetitions. Emphasis is placed on proper knee alignment during exercise. Most of the women exhibit excessive medial rotation and adduction of the femur, resulting in knee valgus. The women will be instructed how to correct their abnormalities using mirrors as visual feedback. All exercises will be completed without pain. If the exercises are too easy, the level of difficulty will be increased individually in accordance with the rehabilitation protocol
  Interventions: Other: Neuromuscular Training
- Shock Wave Therapy (Active Comparator): The ESWT group will will meet the therapist twice in the first week, and once a week after it. ESWT will be applied to the iliotibial band and tensor fascia latae with the following parameters: pressure - 4.5 bar, emission frequency -8 Hz, number of pulses per dose -2,500 per session.
  Interventions: Other: Extracorporeal Shock Wave Therapy (ESWT)

INTERVENTIONS:
Other: Neuromuscular Training — Each session lasted 30 minutes and consisted of three sets of exercises with 20-30 repetitions. Emphasis was placed on proper knee alignment during exercise. Most of the women exhibited excessive medial rotation and adduction of the femur, resulting in knee valgus, although knee varus was also observed. The women were instructed how to correct their abnormalities using mirrors as visual feedback. All exercises were completed without pain. If the exercises were too easy, the level of difficulty was increased individually in accordance with the rehabilitation protocol
  Arms: Neuromuscular Training
Other: Extracorporeal Shock Wave Therapy (ESWT) — ESWT will be applied to the iliotibial band and tensor fascia latae muscle with the following parameters: pressure - 4.5 bar, emission frequency -8 Hz, number of pulses per dose -2,500 per session
  Arms: Shock Wave Therapy

SUMMARY:
The aim of the trial is to compare the efficacy of extracorporeal shock wave therapy (ESWT) versus neuromuscular training (TR) in reducing pain in women with patellofemoral pain (PFP). Women with PFP will be randomly divided into two therapeutic groups: ESWT and TR. The ESWT group will undergo extracorporeal shock wave therapy to the iliotibial band and tensor fascia latae. The TR group will be treated with neuromuscular training. The women's gait will be analysed and the strength of hip abductors and internal rotators will be measured. Additionally, the women's pain and health status will be assessed with the visual analogue scale and the Lysholm Scale. Outcomes will be registered at baseline, and then at five weeks and at three months post-therapy

ELIGIBILITY:
Inclusion Criteria:

Knee pain for more than three months greater than three on the visual analogue scale (VAS) during at least two out of four typical activities:

1. ascending or descending the stairs,
2. prolonged sitting with flexed knee,
3. running or jumping,
4. squatting or kneeling.

Exclusion Criteria:

1. Orthopaedic diagnosis other than PFP.
2. Patients with neurological disorders, history of injury or operations within the symptomatic leg, rheumatoid disease, or pregnancy were also excluded from the study.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-08-01 (Actual); Primary Completion 2018-06-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale is used to assess the subjective Pain. | Outcome measures are obtained at baseline (pre-intervention)
  The participants are asked to make a mark on a 10 cm line that corresponds to the perceived maximal pain, peripatellar or retropatellar, they experienced during any activity or position (0 = no pain, 10 = the worst pain possible)
Visual Analog Scale is used to assess the subjective Pain. | Outcome measures are obtained, at five weeks after intervention.
  The participants are asked to make a mark on a 10 cm line that corresponds to the perceived maximal pain, peripatellar or retropatellar, they experienced during any activity or position (0 = no pain, 10 = the worst pain possible)
Visual Analog Scale is used to assess the subjective Pain. | Outcome measures are obtained at three months after intervention
  The participants are asked to make a mark on a 10 cm line that corresponds to the perceived maximal pain, peripatellar or retropatellar, they experienced during any activity or position (0 = no pain, 10 = the worst pain possible)

SECONDARY OUTCOMES:
Gait analysis using the Zebris FDM-TDL instrumented treadmill with pressure sensors. | Outcome measures are obtained at baseline (pre-intervention)
  The women walk on the treadmill barefoot for three minutes in order to become accustomed to the speed belt. After that time, the angles of the joints are measured for 30 seconds. Internal rotation is demarcated at the highest peak in midstance when the contralateral limb is in the terminal stance (toe-off phase). Hip adduction is determined at the highest peak in midstance
Gait analysis using the Zebris FDM-TDL instrumented treadmill with pressure sensors. | Outcome measures are obtained, at five weeks after intervention.
  The women walk on the treadmill barefoot for three minutes in order to become accustomed to the speed belt. After that time, the angles of the joints are measured for 30 seconds. Internal rotation is demarcated at the highest peak in midstance when the contralateral limb is in the terminal stance (toe-off phase). Hip adduction is determined at the highest peak in midstance
Gait analysis using the Zebris FDM-TDL instrumented treadmill with pressure sensors. | Outcome measures are obtained at three months after intervention
  The women walk on the treadmill barefoot for three minutes in order to become accustomed to the speed belt. After that time, the angles of the joints are measured for 30 seconds. Internal rotation is demarcated at the highest peak in midstance when the contralateral limb is in the terminal stance (toe-off phase). Hip adduction is determined at the highest peak in midstance
Muscle strength is tested using the Micro Fet Handheld Dynamometer. | Outcome measures are obtained at baseline (pre-intervention)
  Muscle strength of lateral rotators, abductors of the hip is tested. Three repetitions of muscle strength testing are performed with two 30-second intervals. The participants a of re asked to press against the Dynamometer with the maximum effort for 5-7 seconds.
Muscle strength is tested using the Micro Fet Handheld Dynamometer. | Outcome measures are obtained, at five weeks after intervention.
  Muscle strength of lateral rotators, abductors of the hip is tested. Three repetitions of muscle strength testing are performed with two 30-second intervals. The participants a of re asked to press against the Dynamometer with the maximum effort for 5-7 seconds.
Muscle strength is tested using the Micro Fet Handheld Dynamometer. | Outcome measures are obtained at three months after intervention
  Muscle strength of lateral rotators, abductors of the hip is tested. Three repetitions of muscle strength testing are performed with two 30-second intervals. The participants a of re asked to press against the Dynamometer with the maximum effort for 5-7 seconds.
The self-reported health status is measured using the Lysholm Questionaire (LQ) | Outcome measures are obtained at baseline (pre-intervention)
  The participants are asked to complete the eight-item questionnaire, scored on a 0-100 weighted scale
The self-reported health status is measured using the Lysholm Questionaire (LQ) | Outcome measures are obtained, at five weeks after intervention.
  The participants are asked to complete the eight-item questionnaire, scored on a 0-100 weighted scale
The self-reported health status is measured using the Lysholm Questionaire (LQ) | Outcome measures are obtained at three months after intervention
  The participants are asked to complete the eight-item questionnaire, scored on a 0-100 weighted scale

CONTACTS AND LOCATIONS:
Overall Officials: Mgdalena Dabrowska-Galas, PhD, Study Chair — Department of Kinesitherapy and Special Methods, SHS in Katowice, Medical University of Silesia, Katowice, Poland
Locations (1):
- Department of Kinesitherapy and Special Methods, SHS in Katowice, Medical University of Silesia, Katowice, Poland, Katowice, Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided
The datasets used and/or analysed during the current study will be available from the corresponding author on reasonable request.